CLINICAL TRIAL: NCT02568878
Title: An Open-Label Pilot Study of Creatine for Depressed Male and Female Methamphetamine Users
Brief Title: Creatine for Depressed Male and Female Methamphetamine Users
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Montana State University (Other)
Responsible Party: Principal Investigator, Tracy Hellem, Assistant Professor, Montana State University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 01
Record Dates: First submitted 2015-10-01; First posted 2015-10-06 (Estimated); Last update posted 2015-12-11 (Estimated); Status verified 2015-12

CONDITIONS: Depression; Anxiety; Methamphetamine Dependence
Keywords: Depression; Anxiety; Methamphetamine dependence
MeSH Terms: conditions — Depression; Anxiety Disorders | interventions — Creatine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Creatine monohydrate (Experimental): 5 grams of daily creatine monohydrate by mouth for 8 weeks
  Interventions: Drug: Creatine monohydrate

INTERVENTIONS:
Drug: Creatine monohydrate
  Other Names: Creapure

SUMMARY:
* Assess the antidepressant/anxiolytic effect of creatine in male and female methamphetamine users
* Assess creatine's effect on methamphetamine use
* Assess the safety of creatine in male methamphetamine users with depression

ELIGIBILITY:
Inclusion Criteria:

* Current primary diagnosis of methamphetamine dependence or abuse, with methamphetamine preferred drug of abuse
* Current diagnosis of major depressive disorder (primary or substance-induced)
* Current diagnosis of an anxiety disorder (primary or substance-induced)
* Current Hamilton Depression Rating scale score > or = to 16
* Current Hamilton Anxiety Scale score > = to 18
* If taking a psychotropic medication for depressed or anxious mood, regimen must be stable for > = to 4 weeks prior to creatine treatment initiation

Exclusion Criteria:

* Persons unable to provide adequate informed consent
* Persons who are at clinically significant suicidal or homicidal risk
* Primary substance-related diagnosis other than methamphetamine dependence or abuse
* Positive pregnancy test (females only)
* History of renal disease
* Clinically significant medical or neurological illness identified by history, physical exam and laboratory testing
* History of hypersensitivity reaction to creatine

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 29 (Estimated)
Dates: Start 2015-11; Primary Completion 2016-10 (Estimated); Study Completion 2017-05 (Estimated)

PRIMARY OUTCOMES:
Hamilton Depression Rating Scale (HAMD) Scores | This data will be assessed after 12 participants have completed the study and again after a completed sample size of 24 is achieved. The data will be presented at study completion (anticipated: 12 months after study initiation).
Hamilton Anxiety Rating Scale (HAMA) Scores | This data will be assessed after 12 participants have completed the study and again after a completed sample size of 24 is achieved. The data will be presented at study completion (anticipated: 12 months after study initiation).

SECONDARY OUTCOMES:
Self-reported methamphetamine use | This data will be assessed after 12 participants have completed the study and again after a completed sample size of 24 is achieved. The data will be presented at study completion (anticipated: 12 months after study initiation).
Incidence of treatment-emergent adverse events | Adverse events will be reviewed monthly for safety concerns and presented at study completed (anticipated: 12 months after study initiation).
Percent of positive urine drug screens for methamphetamine | This data will be assessed after 12 participants have completed the study and again after a completed sample size of 24 is achieved. The data will be presented at study completion (anticipated: 12 months after study initiation).

CONTACTS AND LOCATIONS:
Overall Officials: Tracy Hellem, PhD, Principal Investigator — Montana State University
Locations (1):
- Montana State University College of Nursing (Missoula campus), Missoula, Montana, United States